CLINICAL TRIAL: NCT02538081
Title: Nicotinic Receptors and Schizophrenia
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Withdrawn
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLNA-008-14S; 14-1443 (Other: University of Colorado, Denver)
Record Dates: First submitted 2015-08-10; First posted 2015-09-02 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Schizophrenia
Keywords: schizophrenia; olanzapine; risperidone; alpha 7 nicotinic receptors; cognition
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone; 3-(2,4-dimethoxybenzylidene)anabaseine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Risperidone plus placebo (Active Comparator): Risperidone titrated to a dose equivalency of the patients' prior dose of olanzapine plus placebo
  Interventions: Drug: Risperidone plus Placebo
- Risperidone plus DMXB-A (Active Comparator): Risperidone titrated to a dose equivalency of the patients' prior dose of olanzapine plus DMXB-A
  Interventions: Drug: Risperidone plus DMXB-A

INTERVENTIONS:
Drug: Risperidone plus Placebo — Standard of care including Risperidone plus Placebo
  Other Names: Risperdal
  Arms: Risperidone plus placebo
Drug: Risperidone plus DMXB-A — Standard of care including Risperidone plus DMXB-A
  Other Names: Risperdal
  Arms: Risperidone plus DMXB-A

SUMMARY:
This study proposes to conduct a clinical trial comparison of olanzapine and the combination of a nicotinic cholinergic agonist, 3-[2,4-Dimethoxybenzylidene]anabaseine (DMXB-A) with a dopamine D2 receptor antagonist, the mechanism common to all antipsychotic drugs, to test the hypothesis that 7-nicotinic receptor agonism may be an additional necessary factor that enhances the efficacy of olanzapine that allows its slight superiority to risperidone. This trial would enroll patients taking olanzapine and record baseline measurements of clinical symptoms, cognition, metabolic parameters, and extrapyramidal side effects. The subjects would then be randomized to receive either risperidone or risperidone plus DMXB-A for 6 weeks and then would again have measurements of clinical symptoms, cognition, metabolic parameters and extrapyramidal side effects.

DETAILED DESCRIPTION:
Basic investigations in both animals and humans point to an increase in cholinergic neurotransmission as one possible mechanism of clozapine and olanzapine's enhanced therapeutic effects. However, there has not been a specific clinical trial to determine if stimulation of a nicotinic cholinergic receptor would capture this enhancement and be safer for patients. In the Clinical Antipsychotic Trials of Intervention Effectiveness (CATIE) those assigned to risperidone from olanzapine had significantly higher discontinuation rates, with the primary reason being lack of efficacy. Olanzapine assignment for all patients was associated with continuing weight gain, which was not seen in patients assigned to risperidone. Many patients assigned to olanzapine from risperidone discontinued because of intolerability of the olanzapine, with metabolic problems being the chief reason. Thus, risperidone is a safer drug and, while equally effective for some patients, for others olanzapine continues to be more effective and tolerated despite its metabolic effect. The baseline rates on entry into the study are typical of most surveys of chronically ill patient populations; about twice as many were receiving olanzapine as were receiving risperidone, which suggests that clinicians choose to treat many patients on olanzapine, despite its side effects, because they do not do well on most other antipsychotic drugs.

This study proposes to conduct a clinical trial comparison of olanzapine and the combination of a nicotinic cholinergic agonist, 3-[2,4-Dimethoxybenzylidene]anabaseine (DMXB-A) with a dopamine D2 receptor antagonist, the mechanism common to all antipsychotic drugs, to test the hypothesis that 7-nicotinic receptor agonism may be an additional necessary factor that enhances the efficacy of olanzapine that allows its slight superiority to risperidone. In pilot data, the investigators studied 11 patients who received DMXB-A 300 mg plus olanzapine 20 mg (n=5) or risperidone 4 mg (n=6). The investigators found that DMXB-A improved performance on the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) mean battery score of the risperidone-treated patients to the level of the olanzapine-treated patient.

This trial would enroll patients taking olanzapine and record baseline measurements of clinical symptoms, cognition, metabolic parameters, and extrapyramidal side effects. The subjects would then be randomized to receive either risperidone or risperidone plus DMXB-A for 6 weeks and then would again have measurements of clinical symptoms, cognition, metabolic parameters and extrapyramidal side effects.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 25
* Diagnosis of schizophrenia or schizoaffective disorder
* 18-75 years of age
* Taking olanzapine at least 10 mg
* If female, willing to use acceptable birth control during the study
* fluent in english

Exclusion Criteria:

* No emergent serious medical issues:

  * cardiovascular disease
  * neurological illnesses including -

    * severe head injury
    * HIV infection
    * liver disease
    * blood diseases
    * kidney disease
* No drugs of abuse
* Not pregnant
* Not able to fast
* History of severe head injury

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in Attention due to DMXB-A | measured at 6 weeks
  the difference in the attention index from the RBANS measured at 6 weeks between risperidone plus DMXB-A and risperidone plus placebo
Change in Executive Function due to DMXB-A | measured at 6 weeks
  the difference in the executive function index from the RBANS measured at 6 weeks between risperidone plus DMXB-A and risperidone plus placebo

SECONDARY OUTCOMES:
Change in LDL | measured at 6 weeks
  the difference in LDL at 6 weeks on risperidone plus placebo or risperidone plus DMXB-A
Change in HDL | measured at 6 weeks
  the difference in HDL measured at 6 weeks between risperidone plus placebo and risperidone plus DMXB-A
Change in glucose | measured at 6 weeks
  the difference in glucose measured at 6 weeks on either risperidone plus placebo and risperidone plus DMXB-A
Change in Hemoglobin A1C | measured at 6 weeks
  The difference in hemoglobin A1C measured at 6 weeks on either risperidone plus placebo and risperidone plus DMXB-A
Change in insulin levels | measured at 6 weeks
  The difference in insulin levels measured at 6 weeks between on either risperidone plus placebo and risperidone plus DMXB-A
Change in c-reactive protein | measured at 6 weeks
  The difference in C-reactive protein measured at 6 weeks between risperidone plus placebo and risperidone plus DMXB-A
Change in girth | measured at 6 weeks
  The difference in girth measured at 6 weeks between risperidone plus placebo and risperidone plus DMXB-A
Change in BMI | measured at 6 weeks
  The difference in BMI measured at 6 weeks between risperidone plus placebo and risperidone plus DMXB-A
Change in Cholesterol | measured at 6 weeks
  The difference in Cholesterol measured at 6 weeks between risperidone plus placebo and risperidone plus DMXB-A
Change in the total scale score of the brief psychiatric rating scale | measured at 2 weeks, 3 weeks, 4 weeks, 5 weeks and 6 weeks of drug administration, or, if the subject exits the study prematurely, on the day of study exit.
  The difference in the Total scale score of the Brief Psychiatric Rating Scale BPRS measured at 6 weeks or at study conclusion on either risperidone plus placebo and risperidone plus DMXB-A
Change in the scale for the assessment of negative symptoms | measured at 2 weeks, 3 weeks, 4 weeks, 5 weeks and 6 weeks
  The difference in the clinical Scale for the Measurement of Negative Symptoms (SANS) measured at 6 weeks on either risperidone plus placebo and risperidone plus DMXB-A
Change in Attention index with switch from olanzapine to risperidone plus DMXB-A | measured at baseline and 6 weeks
  The difference in the attention index from the RBANS measured on olanzapine at baseline and at 6 weeks on risperidone plus DMXB-A
Change in Executive function index with switch from olanzapine to risperidone plus DMXB-A | measured at baseline and 6 weeks
  The difference in the executive function index from the RBANS measured on olanzapine at baseline and at 6 weeks on risperidone plus DMXB-A
Change in Total BPRS with switch from olanzapine to risperidone plus DMXB-A | measured at baseline and 6 weeks
  The difference in the Total BPRS measured on olanzapine at baseline and at 6 weeks on risperidone plus DMXB-A
Change in SANS with switch from olanzapine to risperidone plus DMXB-A | measured at baseline and 6 weeks
  The difference in the SANS measured on olanzapine at baseline and at 6 weeks on risperidone plus DMXB-A
Change in BMI with switch from olanzapine to risperidone plus DMXB-A | measured at baseline and 6 weeks
  The difference in the BMI measured on olanzapine at baseline and at 6 weeks on risperidone plus DMXB-A
Change in c-reactive protein with switch from olanzapine to risperidone plus DMXB-A | measured at baseline and 6 weeks
  The difference in the c-reactive protein measured on olanzapine at baseline and at 6 weeks on risperidone plus DMXB-A
Change in LDL with switch from olanzapine to risperidone plus DMXB-A | measured at baseline and 6 weeks
  The difference in the LDL measured on olanzapine at baseline and at 6 weeks on risperidone plus DMXB-A
Change in HDL with switch from olanzapine to risperidone plus DMXB-A | measured at baseline and 6 weeks
  The difference in the HDL measured on olanzapine at baseline and at 6 weeks on risperidone plus DMXB-A
Change in glucose with switch from olanzapine to risperidone plus DMXB-A | measured at baseline and 6 weeks
  The difference in the glucose measured on olanzapine at baseline and at 6 weeks on risperidone plus DMXB-A
Change in cholesterol with switch from olanzapine to risperidone plus DMXB-A | measured at baseline and 6 weeks
  The difference in the cholesterol measured on olanzapine at baseline and at 6 weeks on risperidone plus DMXB-A
Change in cholesterol with switch from olanzapine to risperidone plus DMXB-A | measured at baseline and 6 weeks
  The difference cholesterol measured on olanzapine at baseline and at 6 weeks on risperidone plus DMXB-A
Change in girth with switch from olanzapine to risperidone plus DMXB-A | measured at baseline and 6 weeks
  The difference girth measured on olanzapine at baseline and at 6 weeks on risperidone plus DMXB-A
Change in insulin levels with switch from olanzapine to risperidone plus DMXB-A | measured at baseline and 6 weeks
  The difference insulin levels measured on olanzapine at baseline and at 6 weeks on risperidone plus DMXB-A
Change in hemoglobin A1C with switch from olanzapine to risperidone plus DMXB-A | measured at baseline and 6 weeks
  The difference in Hemoglobin A1C measured on olanzapine at baseline and at 6 weeks on risperidone plus DMXB-A

CONTACTS AND LOCATIONS:
Overall Officials: Robert Freedman, MD, Principal Investigator — VA Eastern Colorado Health Care System, Denver, CO
Locations (1):
- VA Eastern Colorado Health Care System, Denver, CO, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No